CLINICAL TRIAL: NCT05100537
Title: The Effect of Mindfulness Based Stress Reduction Programme for Reducing the Stress Level and Emotion Regulation of Nursing Students
Brief Title: Effect of Mindfulness Based Stress Reduction (MBSR) Programme for Reducing the Stress Level of Nursing Student
Acronym: MBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Ece Alagoz, Lecturer, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0051
Record Dates: First submitted 2021-10-05; First posted 2021-10-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Stress; Emotion Regulation
Keywords: Mindfulness; Nursing student
MeSH Terms: conditions — Emotional Regulation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): The Mindfulness Based Stress Reduction program is a manualized course that includes meditation, relaxing movement, and breathing. A certified MBSR instructor will teach the courses in a group-based format for 120 minute sessions, once per week for eight weeks.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- CONTROL GROUP (Active Comparator): no intervention
  Interventions: Other: continuing a routine life

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — The intervention has its roots in meditations and yoga practices. However, it is independent of religious purpose or affiliation.The weekly sessions include a range of mental and bodily practices, including awareness of emotions, awareness of thoughts, awareness of sensations. It involves full awareness of daily activities, using the breath as an anchor for attention.In addition to mindfulness practices and experiential work, psychoeducation and participants' sharing will clarify the issues of stress, stress management and how mindfulness is applied in daily situations and interpersonal communication.
  Arms: Mindfulness Based Stress Reduction
Other: continuing a routine life — No intervention will be made in the control group.
  Arms: CONTROL GROUP

SUMMARY:
Purpose: This research was planned to determine the effect of mindfulness-based stress reduction program on reducing the stress level and emotion regulation of nursing students.

Design: The research was planned as a pretest, posttest, follow-up and randomized controlled study in order to determine the effect of the mindfulness-based stress reduction program on the stress level and emotion regulation of nursing students.

Hypotheses: H1: The perceived stress level scores of nursing students in the intervention group participating in the mindfulness-based stress reduction program will decrease compared to the nursing students in the control group.

H2: The perceived stress level of the nursing students in the intervention group participating in the mindfulness-based stress reduction program will decrease according to their pretest scores.

H3: Emotion regulation strategies of nursing students in the intervention group participating in the mindfulness-based stress reduction program will differ from the nursing students in the control group.

H4: The posttest and follow-up emotion regulation strategies of nursing students in the intervention group participating in the mindfulness-based stress reduction program will differ from the pretest.

ELIGIBILITY:
Inclusion Criteria:

* Age range is 18-25 years old
* Being a student in the second or third year of the nursing department
* Regular attendance at school
* Not having a communication problem related to vision or hearing
* It was determined as having a score of 26 or more from the perceived stress scale.

Exclusion Criteria:

* Have a psychiatric illness

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | For 3 months
  The 14-item scale was designed to measure how stressful the individual perceives certain situations in his life. The scale is in 5-point Likert type, ranging from "Never (0)" to "Very often (4)". 7 of the scale items with positive expressions are scored in reverse. The total score from the scale indicates the stress level of the person. A score between 11-26 indicates a low stress level, a score between 27-41 indicates a medium stress level, and a score between 42-56 indicates a high stress level.
Cognitive Emotion Regulation Scale | For 3 months
  It is a five-point Likert type scale (1 = not at all suitable for me, 2 = somewhat suitable for me, 3 = somewhat suitable for me, 4 = very suitable for me, 5 = completely suitable for me). The scale consists of 36 items in total. Cronbach's alpha value in the original form of the scale. with 67. It is between 81. The scale includes "self-blame", "acceptance", "focus on thought", "positive refocus", "plan refocus", "positive reconsideration", "perspective", "destruction" and "blaming others". It consists of nine sub-dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ece alagöz, Pendik, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No